CLINICAL TRIAL: NCT06044844
Title: A Study Evaluating the Effectiveness of Tofacitinib in Systemic Sclerosis
Brief Title: Effectiveness of Tofacitinib in Systemic Sclerosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Collaborators: Aristopharma Ltd (Industry)
Responsible Party: Principal Investigator, Nabil Amin Khan, Resident,rheumatology, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4137
Record Dates: First submitted 2023-06-07; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Efficacy of Tofacitinib in the Systemic Sclerosis
MeSH Terms: interventions — tofacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- efficacy of tofacitinib in early diffuse cutaneous systemic sclerosis (Experimental): tab tofacitinib 5mg twice daily will be given by oral route for 6month
  Interventions: Drug: Tofacitinib
- efficacy of Cyclophosphamide in early diffuse cutaneous systemic sclerosis (Experimental): injection cyclophosphamide 500mg/m2 body surface area/monthly by intravenous infusion.total 6cycle will be given
  Interventions: Drug: Tofacitinib

INTERVENTIONS:
Drug: Tofacitinib — tofacitinib efficacy
  Other Names: Tab Arthanib

SUMMARY:
The goal of this clinical trial is to compare efficacy of tofacitinib with cyclophosphamide in skin thickening in early diffuse cutaneous systemic sclerosis .

DETAILED DESCRIPTION:
compare tofacitinib 5mg twice daily with cyclophosphamide 500mg/m2/month in early diffuse cutaneous systemic sclerosis

ELIGIBILITY:
* Inclusion criteria:

  1. Diagnosis of SSc, as classified using the 2013 American College of Rheumatology
  2. dcSSc as defined by 2001 LeRoy and Medsge
  3. Disease duration ≤ 60 months (defined as time from the first non-Raynaud phenomenon manifestation)
  4. mRSS units ≥ 10 and ≤ 45 at screening.
  5. Oral corticosteroids (≤ 10 mg/day of prednisone or equivalent) are permitted if the patient is on a stable dose regimen for ≥ 2 weeks prior to and including the baseline visit.
  6. Calcium channel blocker and PDFE-5 inhibitors for Raynaud's and digital ulcers are permitted to use as oral monotherapy
  7. Age ≥ 18 years and ≤ 70 years
  8. Ability to provide informed consent.

Exclusion Criteria:

Subjects with any of the following characteristics/conditions will not be included in the study:

1. Any infection at screening .
2. Oral corticosteroids >10 mg/day of prednisone or equivalent.
3. Pulmonary disease with FVC ≤ 35% of predicted.
4. Subjects at risk for tuberculosis (TB).Specifically excluded from this study with a history of active TB within the last 3 years and current clinical, radiographic, or laboratory evidence of active TB.j
5. Latent TB at or within 30 days of screening.
6. Positive for hepatitis B surface antigen at or within 30 days of screening.
7. Positive for hepatitis C antigen at or within 30 days of screening.
8. Current or recent history of uncontrolled clinically significant renal, hepatic, hematologic, gastrointestinal, metabolic, endocrine, pulmonary, cardiac or neurologic disease.
9. History of diverticulitis or chronic, ulcerative lower GI disease such as Crohns disease, ulcerative colitis, or other symptomatic, lower GI conditions that might predispose a patient to perforations.
10. Pregnant or breastfeeding female subjects and female subjects of childbearing potential who are unwilling or unable to use a highly effective method of contraception as outlined in the protocol for the duration of the study and for at least 28 days after discontinuation of study drug.
11. History of any malignancy in the last 5 years with the exception of adequately treated or excised basal cell or squamous cell or cervical cancer in situ.
12. History of SSc Renal Crisis within the 6 months prior to baseline.
13. History of live/attenuated vaccine ≤ 6 weeks prior to baseline
14. Any of the following lab results at screening:

    * Hemoglobin <9 g/dL or Hematocrit <30%
    * White Blood Cell count <3.0 x 109/L;
    * Absolute Neutrophil count <1.2 x 109/L;
    * Platelet count <100 x 109/L;
    * Absolute Lymphocyte count <0.75 x 109/L.
    * ALT or AST > 3 × the upper limit of normal (ULN) of normal at screening or any
    * Total bilirubin > ULN at Screening.
    * Estimated glomerular filtration rate [GFR] <40mL/min/1.73 m2

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
skin thickness | 24 weeks after initiation of treatment
  skin thickness measured by modified rodnan skin score

SECONDARY OUTCOMES:
joint pain | 24 weeks after initiation of treatment
  measured by clinical disease activity index

CONTACTS AND LOCATIONS:
Overall Officials: Nabil Khan, MBBS, Principal Investigator — resident
Locations (1):
- Nabil Amin Khan, Dhaka, Shahbag, Bangladesh

IPD SHARING:
Plan to Share IPD: No